CLINICAL TRIAL: NCT05539950
Title: Cardiopulmonary Rehabilitation in Post-acute COVID-19 Syndrome
Acronym: COVID-19
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to get funds
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Hung-Chou Chen, Director and Attending Physician, Taipei Medical University Shuang Ho Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMU-IJRB-N202208050
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Post Acute COVID-19 Syndrome
Keywords: Long COVID; Cardiopulmonary rehabilitation
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiopulmonary rehabilitation with health education (Experimental): The participants will participate in cardiopulmonary rehabilitations programs under the supervision of therapists 3 times a week, 12 weeks in total. Recommendations for individualized exercise prescription and lifestyle modification will be given to the participants as well.
  Interventions: Other: Cardiopulmonary rehabilitation; Other: Health education
- Health education (Active Comparator): The participants will be given recommendations for individualized exercise prescription and lifestyle modification.
  Interventions: Other: Health education

INTERVENTIONS:
Other: Cardiopulmonary rehabilitation — Cardiopulmonary rehabilitation helps patients maximize functional potential due to progressive deconditioning or acute decompensation following an acute medical event. This intervention is medically supervised and individualized according to their results of the cardiopulmonary Exercise Testing (CPET).
  Arms: Cardiopulmonary rehabilitation with health education
Other: Health education — Individualized exercise prescription will be given according to their results of the cardiopulmonary Exercise Testing (CPET). Recommendations for lifestyle modification will also be given.

SUMMARY:
In 2022, though the optimized acute medical treatment of COVID-19 was determined, patients often experience the sequelae (also known as post-acute COVID-19 syndrome, the patients might develop cough, breathlessness, fatigue, weakness, impaired activities of daily livings etc.). Until now, there is no consensus for post-acute COVID-19 syndrome management. Previously, the cardiopulmonary rehabilitation revealed significant benefits in heart failure or chronic obstructive pulmonary disease. The aims of the study are demonstrating the benefits and safety of cardiopulmonary rehabilitations in patients previously admitted to hospital because of COVID-19 with sequelae.

DETAILED DESCRIPTION:
PURPOSE: To demonstrate the benefits and safety of cardiopulmonary rehabilitations in patients previously admitted to hospital because of COVID-19 with sequelae.

METHODS: The participants will be divided into two groups: one with cardiopulmonary rehabilitations programs under the supervision of therapists 3 times a week, 12 weeks in total with lifestyle modification (experimental group); and the other with lifestyle modification and health education (active-controlled group). Before and after the interventions, several endpoints in interested are performed by the physicians or the research assistants, including cardiopulmonary exercise training (CPET), 6-minute-walk-test (6MWT), pulmonary function tests (PFT), and quality of life (QoL, we plan to use SF-36) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* be willing and able to provide written informed consent and comply with all procedures required by the protocol
* be 20 - 80 years of age at the time of signing the Informed Consent Form
* diagnosed with COVID-19 with PCR and admitted with at least moderate COVID-19 disease (with clinical symptoms or imaging evidence of low respiratory tract involvement)
* diagnosed with COVID-19 for over 4 weeks but less than 2 years with fatigue, shortness of breath, cough, weakness, or impairments of activities of daily life
* able to cooperate with the rehabilitation programs and cycling

Exclusion Criteria:

* Patients under 20-year-old or over 80-year-old, pregnant, prisoners
* Patients without national health insurance in Taiwan
* The patient cannot follow instructions or cycling

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Cardiopulmonary exercise testing (CPET) | Baseline, Week 12
  CPET is a non-invasive examination, which provides assessment of the integrative exercise responses involving the pulmonary, cardiovascular, hematopoietic, neuropsychological, and skeletal muscle systems. It permits the evaluation of both submaximal and peak exercise responses. CPET is currently act as a clinical applications for the evaluation of undiagnosed exercise intolerance and for the objective determination of functional capacity and impairment.

SECONDARY OUTCOMES:
Changes in 6 minutes walking test (6MWT) | Baseline, Week 12
  6MWT is a commonly used test for the objective assessment of functional exercise capacity for the management of patients with moderate-to-severe pulmonary disease. This test does not require complex equipment or technical expertise. The participant is asked to walk as far as possible along a 30-m minimally trafficked corridor for a period of 6 min with the primary outcome measure being the 6-min walk distance (6MWD) measured in meters.
Changes in Pulmonary function test (PFT) | Baseline, Week 12
  PFT is used in investigating and monitoring of patients with respiratory pathology. PFT allows physicians to quantify the severity of the pulmonary disease, follow it up over time, and assess its response to treatment.
Changes in 36-Item Short Form Survey (SF-36) | Baseline, Week 12
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. This questionnaire includes one multi-item scale that assesses eight health concepts: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University-Shuang Ho Hospital, Ministry of Health and Welfare, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albouaini K, Egred M, Alahmar A, Wright DJ. Cardiopulmonary exercise testing and its application. Postgrad Med J. 2007 Nov;83(985):675-82. doi: 10.1136/hrt.2007.121558. PMID 17989266
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Agarwala P, Salzman SH. Six-Minute Walk Test: Clinical Role, Technique, Coding, and Reimbursement. Chest. 2020 Mar;157(3):603-611. doi: 10.1016/j.chest.2019.10.014. Epub 2019 Nov 2. PMID 31689414
- [Background] Ponce MC, Sankari A, Sharma S. Pulmonary Function Tests. 2023 Aug 28. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482339/ PMID 29493964